CLINICAL TRIAL: NCT06248814
Title: A Phase 1b, Randomized, Double-blind, Placebo-controlled, Single Dose, Crossover Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of BMS-986326 at Two Dose Levels in Adult Participants With Atopic Dermatitis
Brief Title: A Study to Evaluate the Safety, Tolerability, Drug Levels, and Drug Effects of BMS-986326 in Participants With Atopic Dermatitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IM034-1014; 2022-502997-18 (Registry Identifier: EU Trial Number)
Record Dates: First submitted 2024-01-31; First posted 2024-02-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Dermatitis, Atopic
Keywords: Skin Disease; Dermatitis; Eczema
MeSH Terms: conditions — Dermatitis, Atopic; Skin Diseases; Dermatitis; Eczema

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Placebo, followed by BMS-986326 Dose A or Dose B (Experimental)
  Interventions: Drug: BMS-986326; Other: Placebo
- BMS-986326 Dose A, followed by Placebo (Experimental)
  Interventions: Drug: BMS-986326; Other: Placebo
- BMS-986326 Dose B, followed by Placebo (Experimental)
  Interventions: Drug: BMS-986326; Other: Placebo

INTERVENTIONS:
Drug: BMS-986326 — Specified dose on specified days
Other: Placebo — Specified dose on specified days

SUMMARY:
The purpose of this study is to assess the safety, tolerability, drug levels, drug effects, and impact on disease severity of BMS-986326 in participants with moderate-to-severe atopic dermatitis (AD).

ELIGIBILITY:
Inclusion Criteria:

* Must have diagnosis of atopic dermatitis (AD) at least 12 months prior to screening
* Documented history of inadequate response to treatment with topical medication for at least 4 weeks, unless topical treatments are otherwise medically inadvisable, or has required systemic therapy for control of disease
* All the following must be present to confirm moderate-to-severe AD

  * Eczema Area and Severity Index score ≥ 12 (at Screening and Day 1)
  * Body Surface Area ≥ 10% (at Screening and Day 1)
  * Validated Investigator Global Assessment for Atopic Dermatitis ≥ 3 (at Screening and Day 1)
  * Peak Pruritus Numerical Rating Scale ≥ 4 (at Screening)

Exclusion Criteria:

* Evidence of an active and/or concurrent inflammatory skin condition that would interfere with the Investigator or subject-driven evaluations of AD
* Any major surgery within the last 30 days before the first dose of study intervention, or any surgery planned during the course of the study
* Any other sound medical, psychiatric, and/or social reason as determined by the investigator

Other protocol-defined inclusion/exclusion criteria apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2024-03-06 (Actual); Primary Completion 2025-11-06 (Actual); Study Completion 2025-11-06 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) | Up to approximately 224 days
Number of participants with serious adverse events (SAEs) | Up to approximately 224 days
Number of participants with clinical laboratory abnormalities | Up to approximately 224 days
Number of participants with vital sign abnormalities | Up to approximately 224 days
Number of participants with electrocardiogram (ECG) abnormalities | Up to approximately 224 days
Number of participants with physical examination abnormalities | Up to approximately 224 days

SECONDARY OUTCOMES:
Maximum observed concentration (Cmax) | Up to approximately 224 days
Time of maximum observed concentration (Tmax) | Up to approximately 224 days
Area under the concentration-time curve from time zero to time of last quantifiable concentration [AUC(0-T)] | Up to approximately 224 days
Change from baseline in regulatory T cell (Treg) count | Up to approximately 224 days
Change from baseline in Treg-to- conventional T cell (Tconv) ratio | Up to approximately 224 days
Incidence of anti-drug antibody (ADA) | Up to approximately 224 days
Mean percentage change from baseline at selected visits through 112 days in EASI score | Up to approximately 112 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (13):
- Czechia (2):
  - Local Institution - 0004, Prague, PR
  - Local Institution - 0009, Pardubice
- France (3):
  - Local Institution - 0006, Clermont-Ferrand
  - Local Institution - 0010, Nice
  - Local Institution - 0008, Pierre-Bénite
- Germany (3):
  - Local Institution - 0005, Chemnitz, Saxony
  - Local Institution - 0012, Lübeck, Schleswig-Holstein
  - Local Institution - 0011, Berlin, State of Berlin
- Poland (3):
  - Local Institution - 0015, Krakow, Lesser Poland Voivodeship
  - Local Institution - 0001, Rzeszów, Podkarpackie Voivodeship
  - Local Institution - 0016, Katowice, Silesian Voivodeship
- Spain (2):
  - Local Institution - 0013, Las Palmas de Gran Canaria, GC
  - Local Institution - 0002, Córdoba, X

IPD SHARING:
Plan to Share IPD: No
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosurecommitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSClinicalTrials.com